CLINICAL TRIAL: NCT02694029
Title: Intra-patient Comparison of Active Breathing Coordinator-based vs VisionRT-based Deep Inspiration Breath-hold for Left-chest Wall Irradiation, a Pilot Study for Breast Cancer
Brief Title: Active Breathing Coordinator-based vs VisionRT-based Deep Inspiration Breath-hold for Radiation for Breast Cancer
Acronym: VisionRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Asal Rahimi, ASSOC PROFESSOR, Radiation Oncology - RO-Radiation Oncology, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: STU 052015-047
Record Dates: First submitted 2016-02-11; First posted 2016-02-29 (Estimated); Results first posted 2021-08-06 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ABC (Active Breathing Coordinator ), Then VRT (Active Comparator): Active Breathing Coordinator to assist radiation therapy. This group will be administered 14 fractions with ABC-assisted DIBH, followed by 14 fractions with VRT-assisted DIBH
  Interventions: Device: Active Breathing Coordinator (ABC); Device: VisionRT
- VisionRT (VRT), Then ABC (Active Comparator): VisionRT-based deep inspiration breath-hold to assist radiation therapy. This group will be administered 14 fractions with VRT-assisted DIBH, followed by 14 fractions with ABC-assisted DIBH
  Interventions: Device: Active Breathing Coordinator (ABC); Device: VisionRT

INTERVENTIONS:
Device: Active Breathing Coordinator (ABC) — The ABC system has a digital spirometer that records real time breathing. This group will be administered 14 fractions with ABC-assisted DIBH, followed by 14 fractions with VRT-assisted DIBH
Device: VisionRT — A technology for implementing the deep inspiration breath-hold technique is real-time surface photogrammetry. This group will be administered 14 fractions with VRT-assisted DIBH, followed by 14 fractions with ABC-assisted DIBH.
  Other Names: AlignRT system

SUMMARY:
Female patients treated with radiation for left-sided breast malignancy will undergo alternate fractions of Active Breathing Coordinator (ABC)-assisted and VisionRT-assisted Deep Inspiration Breath-Hold (DIBH).

DETAILED DESCRIPTION:
Female patients treated with radiation for left-sided breast malignancy will undergo alternate fractions of ABC-assisted and VisionRT-assisted DIBH. Residual motion during breath-hold will be quantitatively assessed using MV fluoroscopy from the treatment beam itself (i.e., no additional radiation dose). The dosimetric impact of residual motion on organs at risk (heart and lung) will be assessed by applying rigid and/or deformable displacements to the planning CT images, computing the 3D dose map and comparing with the original planned dose map.

ELIGIBILITY:
Inclusion Criteria:

* Women with diagnosis of breast malignancy
* Women whom requires left chest wall post-mastectomy radiation with or without bolus
* Age ≥ 18 years.
* Performance status ECOG </=3
* Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately Ability to understand and the willingness to sign a written informed consent.
* Patient must be able to maintain a 30 second breath hold.
* Conventional chest wall radiation delivery dose of 50.4 Gy/ 28 fractions with or without a boost (boost will not be evaluated for endpoints)

Exclusion Criteria:

* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Subjects must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-09-04 (Actual); Study Completion 2018-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Asal Rahimi, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- The University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Out of 11 participants consented, 1 participant withdrew before randomization
Groups:
- Arm 1: ABC, Then VRT: Active Breathing Coordinator to assist radiation therapy. This group will be administered 14 fractions with ABC-assisted DIBH, followed by 14 fractions with VRT-assisted DIBH
  Active Breathing Coordinator (ABC): The ABC system has a digital spirometer that records real time breathing. This group will be administered 14 fractions with ABC-assisted DIBH, followed by 14 fractions with VRT-assisted DIBH
- Arm 2: VRT, Then ABC: VisionRT-based deep inspiration breath-hold to assist radiation therapy. This group will be administered 14 fractions with VRT-assisted DIBH, followed by 14 fractions with ABC-assisted DIBH
  VisionRT: A technology for implementing the deep inspiration breath-hold technique is real-time surface photogrammetry. This group will be administered 14 fractions with VRT-assisted DIBH, followed by 14 fractions with ABC-assisted DIBH.
Period: Overall Study
Arm/Group | Arm 1: ABC, Then VRT | Arm 2: VRT, Then ABC
Started | 5 | 5
First Intervention | 5 | 5
Second Intervention | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Breast cancer patients undergoing radiation.
Groups:
- Arm 2: VisionRT, Then ABC: VisionRT-based deep inspiration breath-hold to assist radiation therapy. This group will be administered 14 fractions with VRT-assisted DIBH, followed by 14 fractions with ABC-assisted DIBH
  VisionRT: A technology for implementing the deep inspiration breath-hold technique is real-time surface photogrammetry. This group will be administered 14 fractions with VRT-assisted DIBH, followed by 14 fractions with ABC-assisted DIBH.
- Total: Total of all reporting groups
Arm/Group | Arm 1: ABC, Then VRT | Arm 2: VisionRT, Then ABC | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 8
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 4 | 4 | 8
  Black or African American | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Residual Motion During Deep Inspiratory Breath-Hold (DIBH)
Description: Residual motion is measured as range of breast/chest wall motion during the ABC or VisionRT assisted DIBH beam delivery. The range of motion will be measured in a unit of millimeter.
Time Frame: All patients received treatment for 2 hours for a minimum of 6 weeks
Measure: Mean (Full Range); unit: mm
Groups:
- Radiation With ABC: Active Breathing Coordinator to assist radiation therapy. This group will be administered 14 fractions with ABC-assisted DIBH
  Active Breathing Coordinator (ABC): The ABC system has a digital spirometer that records real time breathing. This group will be administered 14 fractions with ABC-assisted DIBH
- Radiation VRT: VisionRT-based deep inspiration breath-hold to assist radiation therapy. This group will be administered 14 fractions with VRT-assisted DIBH
  VisionRT: A technology for implementing the deep inspiration breath-hold technique is real-time surface photogrammetry. This group will be administered 14 fractions with VRT-assisted DIBH
Arm/Group | Radiation With ABC | Radiation VRT
Number analyzed (Participants) | 10 | 10
mm | 0.27 [-3.0 to 3.1] | 0.27 [-1.8 to 1.8]

2. Secondary Outcome: Time of Simulation
Description: To compare time of simulation and daily treatment for DIBH with both ABC and Vision RT
Time Frame: All patients received treatment for 2 hours for a minimum of 6 weeks
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Radiation With VRT: VisionRT-based deep inspiration breath-hold to assist radiation therapy. This group will be administered 14 fractions with VRT-assisted DIBH
  VisionRT: A technology for implementing the deep inspiration breath-hold technique is real-time surface photogrammetry. This group will be administered 14 fractions with VRT-assisted DIBH
Arm/Group | Radiation With ABC | Radiation With VRT
Number analyzed (Participants) | 10 | 10
minutes | 40.0 (8) | 29.8 (11.4)

3. Secondary Outcome: Time of Treatment in Minutes
Description: To compare time of simulation and daily treatment for DIBH with both ABC and Vision RT
Time Frame: All patients received treatment for 2 hours for a minimum of 6 weeks
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Radiation With ABC: Active Breathing Coordinator to assist radiation therapy. This group will be administered 14 fractions with ABC-assisted DIBH,
  Active Breathing Coordinator (ABC): The ABC system has a digital spirometer that records real time breathing. This group will be administered 14 fractions with ABC-assisted DIBH
- Radiation With VisionRT: VisionRT-based deep inspiration breath-hold to assist radiation therapy. This group will be administered 14 fractions with VRT-assisted DIBH,
  VisionRT: A technology for implementing the deep inspiration breath-hold technique is real-time surface photogrammetry. This group will be administered 14 fractions with VRT-assisted DIBH
Arm/Group | Radiation With ABC | Radiation With VisionRT
Number analyzed (Participants) | 10 | 10
minutes | 9.9 (3.7) | 9.7 (3.8)

4. Secondary Outcome: Reproducibility as Measure of Absolute Change of Breathing Chest Wall Excursion
Description: Reproducibility is defined as the repeatability of inter and intra-fraction DIBH levels. Reproducibility as measure of absolute change of breathing chest wall excursion
Time Frame: All patients received treatment for 2 hours for a minimum of 6 weeks
Measure: Mean (Full Range); unit: mm
Groups:
- Radiation With VisionRT: VisionRT-based deep inspiration breath-hold to assist radiation therapy. This group will be administered 14 fractions with VRT-assisted DIBH
  VisionRT: A technology for implementing the deep inspiration breath-hold technique is real-time surface photogrammetry. This group will be administered 14 fractions with VRT-assisted DIBH
Arm/Group | Radiation With ABC | Radiation With VisionRT
Number analyzed (Participants) | 10 | 10
mm | 0.51 [-11.1 to 8.5] | 0.54 [-5.9 to 8.8]

5. Secondary Outcome: Radiation Dose to Heart
Description: The dosimetric impact of residual motion on heart will be assessed by measuring the radiation dose to heart. We will measure radiation dose by applying rigid displacement to the planing CT and comparing with the original planned dose map.
Time Frame: All patients received treatment for 2 hours for a minimum of 6 weeks
Measure: Mean (Standard Deviation); unit: GY
Arm/Group | Radiation With ABC | Radiation With VRT
Number analyzed (Participants) | 10 | 10
GY | 1.6 (0.7) | 1.6 (0.7)

6. Secondary Outcome: Radiation Dose to Lung
Description: The dosimetric impact of residual motion on lung will be assessed by measuring the radiation dose to lung. We will measure radiation dose by applying rigid displacement to the planing CT and comparing with the original planned dose map.
Time Frame: All patients received treatment for 2 hours for a minimum of 6 weeks
Measure: Mean (Standard Deviation); unit: GY
Arm/Group | Radiation With ABC | Radiation With VisionRT
Number analyzed (Participants) | 10 | 10
GY | 6.3 (1.4) | 6.3 (1.4)

ADVERSE EVENTS:
Time Frame: 30 days
Description: Adverse events were reviewed by treating physicians throughout the treatment duration through standard assessments.
Groups:
- Radiation With ABC: Active Breathing Coordinator to assist radiation therapy. This group will be administered 14 fractions with ABC-assisted DIBH, followed by 14 fractions with VRT-assisted DIBH
  Active Breathing Coordinator (ABC): The ABC system has a digital spirometer that records real time breathing. This group will be administered 14 fractions with ABC-assisted DIBH, followed by 14 fractions with VRT-assisted DIBH
- Radiation With VisionRT: VisionRT-based deep inspiration breath-hold to assist radiation therapy. This group will be administered 14 fractions with VRT-assisted DIBH, followed by 14 fractions with ABC-assisted DIBH
  VisionRT: A technology for implementing the deep inspiration breath-hold technique is real-time surface photogrammetry. This group will be administered 14 fractions with VRT-assisted DIBH, followed by 14 fractions with ABC-assisted DIBH.
Arm/Group | Radiation With ABC | Radiation With VisionRT
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-03): https://cdn.clinicaltrials.gov/large-docs/29/NCT02694029/Prot_SAP_000.pdf